CLINICAL TRIAL: NCT03494543
Title: Endoscopic Papillectomy for Ampullary Adenomas: an Italian Single Centre Experience
Brief Title: Endoscopic Papillectomy for Ampullary Adenomas
Acronym: Papillectomy
Status: Completed | Type: Observational
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Other Study IDs: CORE001
Record Dates: First submitted 2018-04-04; First posted 2018-04-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2018-04

CONDITIONS: Ampullary Adenoma; Familial Adenomatous Polyposis
Keywords: Ampullary Adenoma; Endoscopic Papillectomy; Familial Adenomatous Polyposis
MeSH Terms: conditions — Adenomatous Polyposis Coli

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Endoscopic Papillectomy — Endoscopic resection of ampullary of Vater neoplasms

SUMMARY:
In this single-center experience we retrospectively evaluated principal clinical outcomes of endoscopic papillectomy in all patients referred to our unit. The same evaluation was then performed dividing sproradic ampullary adenoma from familial adenomatous polyposis associated adenomas, and resulting outcomes were compared.

DETAILED DESCRIPTION:
INTRODUCTION Ampullary adenomas are rare tumors of digestive tract with a prevalence of 0.04% to 0.12%, but represent a large part of small intestinal neoplasms. They can origin from the duodenal epithelium or from the pancretobiliary one; the latter seems to have a worse prognosis in terms of nodal metastasis and local invasion with lower long term survival. In these kinds of lesion the adenoma-to-carcinoma sequence has been demonstrated, as already described in the colon.

Symptoms are variable and often are due to the growth of the lesion that can cause pancreatico-biliary obstruction, leading to jaundice and pancreatitis, gastric outlet obstruction, leading to sub-occlusive syndrome or nonspecific abdominal pain, and, rarely, bleeding. Commonly ampullary adenomas are asymptomatic and are discovered during esophagogastroduodenoscopy performed for several symptoms, such as dyspepsia and reflux syndrome, or during endoscopic screening in patients with familial adenomatous polyposis (FAP).

FAP is an autosomal dominant disease caused by mutation in the adenomatous polyposis coli (APC) genes. FAP patients develop colonic polyps in over 90% by age 35 years, while the duodenum is the second most common site of polyp formation. Duodenal/ampullary cancer is the second cause of cancer death in FAP and the risk of development it is 100- to 300-fold higher than the general population and is measured with the Spigelman score that ranges between stage I and IV on the basis of duodenal polyp number, size, histology and grade of dysplasia.

Considering the malignant potential of these lesions, above all in sporadic ampullary adenomas (SAA), complete excision is indicated. Otherwise, in patients with FAP the risk of adenoma to adenocarcinoma transformation seems to be lower and the need of resection is controversial. In the other hand management with annual or biennial surveillance, because of the documented stability of the situation, is suggested only in FAP patients when just minimal irregularity of the papilla is found and low-grade dysplasia was detected.

In the past years pancreatoduodenectomy or transduodenal resection, on the basis of the local invasion and of the local expertise, were the standard treatment, but these approach were burdened by high mortality and morbidity rates. In the last years case reports, retrospective and prospective series have demonstrated the feasibility and safety of the endoscopic resection for benign ampullary adenoma and for early stage ampullary carcinoma with not only diagnostic but also curative intent. Success rate of the endoscopic papillectomy (EP) ranges from 46 to 92% and recurrence rate from 0 to 33% and, recently, the same efficacy with low morbidity respect of surgery have been reported.

In this single-center experience we retrospectively evaluated principal clinical outcomes of EP in all patients referred to our unit. Subsequently the same evaluation was performed dividing SAA from FAP associated adenomas, and resulting outcomes were compared.

METHODS This study is a retrospective analysis of a prospectively collected database. All consecutive patients who underwent EP because of ampullary tumor at Arcispedale Santa Maria Nuova (Reggio Emilia, Italy) between January 2001 and December 2015 were considered. Patients with diagnosis of ampullary adenoma on the endoscopic resection specimen and with at least 24 months of follow-up were included in the analysis. Therefore, patients that underwent EP but without a diagnosis of adenoma or adenocarcinoma in the specimen were excluded from the study.

For all patients preprocedural, procedural and postprocedural data were collected. Preprocedural data were: age, gender, size of the ampullary adenoma, clinical presentation, histology of preprocedural biopsy, endoscopic ultrasound evaluation, and finally, only among patients with FAP, the Spigelman score was calculated. Procedural data were: pancreatic stent placement, biliary stent placement, intraductal invasion. Postprocedural data were: histology of the endoscopic resection specimen and histological subtype, 'en bloc' resection, complete resection, number of procedure to achieve a complete resection, adverse events, need for surgery, recurrence, histology of recurrence, management of recurrence, follow-up and survival.

All patients provided written informed consent to EP. This retrospective study was approved by our Institutional Reviewer Board and, thereafter, by the Ethics Committee.

OUTCOMES The primary outcome of the study was the technical success of EP, considered as achieved when all the following criteria were met: a) complete removal, even in multiple sessions b) absence of residues at histology (histology <= pT1) at the first follow-up; c) recurrence successful treated by endoscopy (not surgery). Technical failure of EP was considered when at least one of the following criteria was met: a) histology> pT1; b) residual adenomatous tissue not suitable of endoscopic resection; c) recurrence treated by surgery. Secondary outcomes were the number of procedures to achieve technical success, the incidence of adverse events, the incidence of recurrence, the concordance of histology pre- and post EP and the evaluation of factors related with technical success.

Finally outcomes of patients with SAA and patients with FAP were compared.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of ampullary adenoma on the endoscopic resection specimen and with at least 24 months of follow-up were included in the analysis

Exclusion Criteria:

* Patients taht underwent endoscopic papillectomy without a diagnosis of adenoma or adenocarcinoma in the specimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who underwent endoscopi papillectomy because of ampullary tumor at Arcispedale Santa Maria Nuova
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
technical success | 24 months
  The primary outcome of the study was the technical success of endoscopic papillectomy, considered as achieved when all the following criteria were met: a) complete removal, even in multiple sessions b) absence of residues at histology (histology <= pT1) at the first follow-up; c) recurrence successful treated by endoscopy (not surgery). Technical failure of EP was considered when at least one of the following criteria was met: a) histology> pT1; b) residual adenomatous tissue not suitable of endoscopic resection; c) recurrence treated by surgery

SECONDARY OUTCOMES:
number of procedures to achieve technical success | 24 months
  number of procedures to achieve technical success
incidence of adverse events | 24 months
  incidence of adverse events
incidence of recurrence | 24 months
  incidence of recurrence
concordance of histology pre- and post endoscopi papillectomy | 24 months
  concordance of histology pre- and post endoscopi papillectomy

CONTACTS AND LOCATIONS:
Overall Officials: Romano Sassatelli, MD, Study Chair — Azienda USL Reggio Emilia - IRCCS

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cecinato P, Parmeggiani F, Braglia L, Carlinfante G, Zecchini R, Decembrino F, Iori V, Sereni G, Tioli C, Cavina M, Camellini L, Azzolini F, Ponz de Leon M, Sassatelli R. Endoscopic Papillectomy for Ampullary Adenomas: Different Outcomes in Sporadic Tumors and Those Associated with Familial Adenomatous Polyposis. J Gastrointest Surg. 2021 Feb;25(2):457-466. doi: 10.1007/s11605-019-04500-w. Epub 2020 Jan 2. PMID 31898110